CLINICAL TRIAL: NCT06511986
Title: Impact of Mechanical Insufflation-Exsufflation on Ventilator-Associated Pneumonia in Post-Neurosurgical Patients: a Safety and Efficacy Study
Brief Title: M-I/E for Preventing VAP in Post-neurosurgical Patients
Status: Completed | Type: Observational
Sponsor: Beijing Sanbo Brain Hospital (Other)
Responsible Party: Principal Investigator, Zhonghua Shi, MD, PhD, vice president of dept. ICU, Beijing Sanbo Brain Hospital
Other Study IDs: VAP prevention
Record Dates: First submitted 2024-07-14; First posted 2024-07-22 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2024-07

CONDITIONS: Ventilator Associated Pneumonia; Brain Injuries; Mechanical Insufflation-exsufflation
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Brain Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Ventilator-associated pneumonia (VAP) is a common infection in critically ill patients, especially those with acute brain injuries, leading to increased mortality and longer ICU stays.

The mechanical insufflation/exsufflation (M-I/E) cough assist device improves outcomes in patients with neuromuscular disorders but its effects on brain-injured patients are largely unknown.

This study is conducted at a tertiary neurosurgical medical center and consists of two substudies. The prospective physiological study assessed the impact of M-I/E on hemodynamics and ICP in mechanically ventilated neurosurgical patients. The combined retrospective-prospective clinical study was performed to investigate the efficacy of M-I/E on occurence of VAP and other clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Post-neurosurgical adult patients
* >18years old
* Body mass index (BMI) <35kg/m2)
* Receiving mechanical ventilation
* With arterial blood catheter for continuous pressure measurement and/or ventricular catheter drainage for ICP measurement (only for study one)

Exclusion Criteria:

* ICP > 22cmH2O or evidence of increased ICP
* Hemodynamically unstable (SBP< 90 or > 160 mmHg; DBP < 50 or > 110 mmHg, using cardiovascular medicine to maintain pressure, or known cardiac failure)
* Patients with lung trauma, emphysema, bronchopleural fistula or risk of pneumothorax
* History of mechanical ventilation and pneumonia within 6 months before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-neurosurgical adult patients receiving mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-01-22 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure | during the process of physiological study, up to 2 hours
  In study one, mean blood pressure will be recorded during the incremental pressure changes in the study one
Heart rate | During the process of physiological study, up to 2 hours
  In study one, heart rate will be recorded during the incremental pressure changes in the study one
Rate of ventilator associated pneumonia | Within 7 days after the onset of mechanical of ventilation
  In study two, ventilator associated pneumonia is defined as pneumonia occurring in patients who have been mechanically ventilated for at least 48 hours. Pneumonia was diagnosed by clinical features (e.g., cough, fever, pleuritic chest pain) and by lung imaging. To derived the diagnosis of pneumonia, patient electronical record, lab results, and images were extracted from the electronical system.

SECONDARY OUTCOMES:
Intracranial pressure | During the process of physiological study, up to 2 hours
  In study one, intracranial pressure will be recorded during the incremental pressure changes in the study one
Length of stay in ICU | Patients will be followed up until 28 days after surgery, discharged from hospital or dead, which ever came first,through study completion, an average of 1 year
  Days of ICU Stay
Length of hospital stay | Patients will be followed up until 28 days after surgery, discharged from hospital or dead, which ever came firstthrough study completion, an average of 1 year
  Days of hospital stay
Days of receiving mechanical ventilation | Patients will be followed up until 28 days after surgery, discharged from hospital or dead, which ever came firstthrough study completion, an average of 1 year
  The duration from the start of mechanical ventilation to the weaning off from ventilator

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Shi, PhD,MD, Principal Investigator — Capital Medical University
Locations (1):
- Beijing Sanbo Brain Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No